CLINICAL TRIAL: NCT01253395
Title: Randomized Equivalency Trial of Strength Compared to Aerobic Exercise on Pain Severity in Adults With Fibromyalgia
Brief Title: Exercise for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: W. Michael Hooten, Md, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005-4167
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Fibromyalgia
Keywords: Exercise; Pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength training (Experimental): Supervised strength training.
  Interventions: Behavioral: Strength training
- Aerobic exercise (Active Comparator): Supervised aerobic exercise.
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Strength training — Daily supervised strength training.
  Arms: Strength training
Behavioral: Aerobic exercise — Daily supervised aerobic exercise.
  Arms: Aerobic exercise

SUMMARY:
Randomized equivalency trial of the effects of strength training compared to aerobic exercise on pain severity in adults with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

- Established diagnosis of fibromyalgia, age > 18 years. Exclusion Criteria: cardiac, pulmonary or orthopedic condition that would limit exercise.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Pain severity | Week 3
  Validated measure of clinical pain.

SECONDARY OUTCOMES:
Muscle strength | Week 3
  Assessment of muscle strength using a dynometer.

CONTACTS AND LOCATIONS:
Overall Officials: William M Hooten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hooten WM, Rosenberg CJ, Eldrige JS, Qu W. Knee extensor strength is associated with pressure pain thresholds in adults with fibromyalgia. PLoS One. 2013;8(4):e59930. doi: 10.1371/journal.pone.0059930. Epub 2013 Apr 2. PMID 23565175
- [Derived] Hooten MW, Qu W, Townsend CO, Judd JW. Effects of strength vs aerobic exercise on pain severity in adults with fibromyalgia: a randomized equivalence trial. Pain. 2012 Apr;153(4):915-923. doi: 10.1016/j.pain.2012.01.020. Epub 2012 Feb 15. PMID 22341565